CLINICAL TRIAL: NCT05603052
Title: A Phase III, Randomized, Observer-blind, Active-controlled, Parallel-group, Multi-center Study to Evaluate Immunogenicity and Safety of a Preventive COVID-19 Vaccine EuCorVac-19 in Healthy Adults Aged 18 Years and Older
Brief Title: A Phase III of COVID-19 Vaccine EuCorVac-19 in Healthy Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EuSNAP_COV302
Record Dates: First submitted 2022-11-01; First posted 2022-11-02 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Test group(EuCorVac-19) - Cohort A (Experimental): Cohort A - Immunogenicity cohort
  Interventions: Biological: EuCorVac-19
- Comparator group(ChAdOx1) - Cohort A (Active Comparator): Cohort A - Immunogenicity cohort
  Interventions: Biological: ChAdOx1 nCoV-19
- Test group(EuCorVac-19) - Cohort B (Experimental): Cohort B - Safety cohort
  Interventions: Biological: EuCorVac-19
- Comparator group(ChAdOx1) - Cohort B (Active Comparator): Cohort B - Safety cohort
  Interventions: Biological: ChAdOx1 nCoV-19

INTERVENTIONS:
Biological: EuCorVac-19 — COVID-19 vaccine
  Arms: Test group(EuCorVac-19) - Cohort A; Test group(EuCorVac-19) - Cohort B
Biological: ChAdOx1 nCoV-19 — COVID-19 vaccine
  Other Names: COVISHIELD
  Arms: Comparator group(ChAdOx1) - Cohort A; Comparator group(ChAdOx1) - Cohort B

SUMMARY:
A phase III, randomized, observer-blind, active-controlled, parallel-group, multi-center study to evaluate immunogenicity and safety of a preventive COVID-19 vaccine EuCorVac-19 in healthy adults aged 18 years and older

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and older who voluntarily decide to participate in this study and provide written informed consent
* Female of childbearing potential who agree to use medically allowed methods of contraception during the study period
* Individuals who agrees not to perform blood donation and transfusion during the study period

Exclusion Criteria:

* Individual being considered to be confirmed COVID-19
* Direct contact with COVID-19 infected person within 14 days prior to the 1st dose of the IP
* Individuals at high risk of exposure to SARS-CoV-2
* Individuals with clinically significant abnormalities in clinical laboratory tests, ECGs, and chest X-ray during screening
* Individuals with fever within 72 hours prior to the 1st dose of the IP or suspected other infectious disease or symptoms associated with other infectious disease
* Individuals with serious medical or psychiatric disease
* History of SARS-CoV or MERS-CoV infection
* History of allergic reaction or hypersensitivity reactions to any of components of the IP
* History of serious adverse events, serious allergic reaction or serious hypersensitivity reactions to vaccination
* History of receiving organ or bone marrow transplant
* Suspected or history of drug abuse or alcohol abuse within 6 months prior to vaccination
* History of vaccination against SARS-CoV, MERS-CoV, or SARS-CoV-2
* History of vaccination with test vaccine substance
* Treatment with immunosuppressants or immune modifying drugs
* History of treatment with antipsychotics or opioid dependence
* Pregnant or lactating women
* Other reasons based on which the individual is considered to be ineligible for this study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2852 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
The proportion of GMT of neutralizing antibody of EuCorVac-19 and ChAdOx1 | 14 days after the 2nd vaccination
The difference in neutralizing antibody SRR of EuCorVac-19 and ChAdOx1 | 14 days after the 2nd vaccination

SECONDARY OUTCOMES:
Occurrence of solicited Adverse Events (AEs) | Through 7 days after each vaccination
Occurrence of unsolicited Adverse Events (AEs) | Through 28 days after the 2nd vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Trial site, Kinshasa, Democratic Republic of the Congo